CLINICAL TRIAL: NCT00687414
Title: Evaluation of Formin Gene Status and Expression in Myeloproliferative and Myelodysplastic Disorders
Status: Completed | Type: Observational
Sponsor: Corewell Health West (Other)
Collaborators: Van Andel Research Institute (Other); Community Foundation for Southeast Michigan (JP McCarthy Fund) (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2008-054
Record Dates: First submitted 2008-05-27; First posted 2008-05-30 (Estimated); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: Myeloproliferative Disorder; MDS; AML
Keywords: gene expression; gene sequencing; gene encoding; MPD; MDS; AML; mDia
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- adults: male and female with MDS and MPD and AML
- Healthy: Healthy control group

SUMMARY:
Aim of the study is to analyze the expression of genes and sequences encoding the human mammalian diaphanous (mDia) related formin proteins to test the hypothesis that defects in the mDia expression or function might drive the pathophysiology of myelodysplastic syndrome, acute myeloid leukemia and other myeloproliferative diseases.

DETAILED DESCRIPTION:
Leukocytes and myeloid lineage cells from these specimens will be assayed for expression of DRF genes using standard molecular biological approaches to measure mRNA levels. Extracted DNA will be analyzed for mutations that affect expressions or function using direct sequencing techniques.

Alternatively, expression of DRF gene products (mDia proteins) will be assessed using specific antibodies and flow cytometry. Molecular findings resulting from these assays will be correlated with clinical information recorded in specimen logbook.

ELIGIBILITY:
Inclusion Criteria:

* 18 and over
* Male
* Female
* Diagnosed with MDS, MPD and AML

Exclusion Criteria:

* Under the age of 18
* Received bone marrow transplant

Control Group Criteria:

inclusion:

* healthy men and women
* ≥ 55 years of age

exclusion:

* history of hematological condition
* history of cancer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Community sample
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2009-12 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
to determine if defective DRF1 expression or mDia1 function may contribute to myeloid malignancies and point to mDia1 as an attractive therapeutic target in MDS and MPS | within a year

CONTACTS AND LOCATIONS:
Overall Officials: Arthur S Alberts, PhD, Principal Investigator — Van Andel Research Institute
Locations (2):
- United States (2):
  - St Mary's Health Care, Grand Rapids, Michigan
  - Van Andel Research Institute, Grand Rapids, Michigan